CLINICAL TRIAL: NCT00000896
Title: A Randomized Controlled Trial to Compare the Efficacy of a Four Drug Antiretroviral Regimen Alone or in Combination With GM-CSF or IL-12 Administered to HIV-1 Infected Subjects as Measured by the Characteristics of Viral Decay
Brief Title: A Study to Compare the Effectiveness of a Four Drug Anti-HIV Regimen Given Alone or in Combination With GM-CSF or IL-12 to HIV-Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 387; 11346 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine; Nevirapine; Stavudine; HIV Protease Inhibitors; Lamivudine; Indinavir; Interleukin-12; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Indinavir; lamivudine, zidovudine drug combination; Hepatitis A Vaccines; Interleukin-12; Nevirapine; Stavudine; sargramostim

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Biological: Hepatitis A Vaccine (Inactivated)
Drug: Interleukin-12
Drug: Nevirapine
Drug: Stavudine
Drug: Sargramostim

SUMMARY:
The purpose of this study is to examine how the level of HIV is reduced in the blood when anti-HIV therapy is initiated. This study will also evaluate whether adding GM-CSF or IL-12 to the anti-HIV drug regimen will increase the rate that HIV is reduced.

The anti-HIV drugs used in this study will include lamivudine (3TC), zidovudine (ZDV), indinavir (IDV), nevirapine (NVP), and stavudine (d4T). All have been used successfully to treat HIV. GM-CSF has been used to treat certain blood disorders; it will be used as an experimental drug in this study. IL-12 (interleukin-12) is a protein found naturally in the body that is thought to boost the immune system. Although GM-CSF and IL-12 have no direct effect against HIV, these drugs may improve the ability of the immune system to fight the virus.

DETAILED DESCRIPTION:
Potent antiretroviral therapies that suppress HIV replication have permitted mathematical modeling of the dynamics of HIV infection and clearance by measurement of the decay of viral load in plasma. When de nova infection is blocked by antiretroviral therapy, the viral load decreases exponentially after a short initial lag time ("shoulder"). This rapid decline is followed by a slower second-phase decay. The intent of this study is to utilize four antiretroviral agents (zidovudine, lamivudine, nevirapine, indinavir) and very frequent measures of viral load to explore the drug-specific kinetics of the "shoulder". The decay of long-lived HIV-infected tissue macrophages is thought to be the major determinant of the slow second phase. Further, the study intends to use immune modulating agents with the potential to increase the turnover of infected macrophages, GM-CSF or IL-12, to accelerate the second phase of viral decay.

Patients are assigned to Group A (16 patients) or to Group B (8 patients). Patients in Group A are randomized to 1 of the following 4 initial treatment arms:

ARM A: Final dose combination (FDC) Zidovudine (ZDV)/Lamivudine (3TC). ARM B: Nevirapine (NVP). ARM C: Indinavir (IDV). ARM D: FDC ZDV/3TC plus NVP plus IDV. The initial regimen is maintained over the first 72 hours and blood for viral dynamic evaluations collected while patients are maintained as inpatients. Then, patients in Arms A, B, and C initiate FDC ZDV/3TC plus NVP plus IDV.

Patients assigned to Group B begin the following 4-drug regimen on Day 0:

ARM E: FDC ZDV/3TC plus NVP plus IDV.

On Day 7, patients in both Groups A and B are randomized to receive one of the following therapies in addition to their 4-drug regimen:

ARM F: GM-CSF daily for 2 weeks, then thrice weekly (MWF). ARM G: IL-12 twice weekly. ARM H: No immune modulation. Patients may be hospitalized to initiate immune modulation or may be treated as outpatients. Immune modulation is discontinued after Week 14. Patients maintain their 4-drug regimen through Week 48. [AS PER AMENDMENT 6/11/99: The study duration has been extended to 96 weeks.] Hepatitis A vaccine (inactivated) is administered on Weeks 16 and 40 [AS PER AMENDMENT 2/13/98: to patients whose baseline hepatitis A serology was negative].

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 cell count greater than or equal to 300 cells/ml within 30 days prior to study entry.
* Have a plasma viral load (level of HIV in the blood) of greater than or equal to 20,000 copies/ml within 30 days of study entry.
* Are at least 18 years old.
* Agree to practice abstinence or use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken anti-HIV medication for more than 7 days.
* Have had known seroconversion within 6 months prior to study entry.
* Have any infection requiring treatment within 30 days prior to study entry.
* Have had a fever for 7 days in a row during the 30 days before study entry.
* Have cancer that requires chemotherapy.
* Are pregnant or breast-feeding.
* Are taking certain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda G. Kost, Study Chair; David Ho, Study Chair
Locations (3):
- United States (3):
  - Ucsd, Avrc Crs, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana